CLINICAL TRIAL: NCT04526730
Title: Neoadjuvant Immunotherapy With Intratumoral Tavokinogene Telseplasmid (Tavo) Plus Electroporation in Combination With Intravenous Nivolumab in Patients With Operable Locally- Regionally Advanced Melanoma
Brief Title: Neoadjuvant Immunotherapy With Tavo + Electroporation in Combination With Nivo. in Melanoma Patients
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: OncoSec Medical Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-20313
Record Dates: First submitted 2020-08-21; First posted 2020-08-26 (Actual); Results first posted 2025-05-06 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Melanoma
Keywords: Skin Cancer
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — Nivolumab; Electroporation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant Treatment (Experimental): Neoadjuvant Phase: (3 x 4-week cycles, total 12 weeks): At every cycle, intratumoral tavo-EP will be administered (on Days 1 and 8) concurrently with 480 mg nivolumab IV infusion on Day 8 of each cycle (tavo-EP will be administered prior to nivolumab infusion).
  Definitive Surgery Phase: Surgery may be scheduled about 2-4 weeks after the last dose of nivolumab following radiologic and clinical assessment at that point. Pathologic response will be determined by institutional pathologist.
  Adjuvant Phase: Adjuvant therapy with nivolumab monotherapy will begin approximately 2-4 weeks following definitive surgery; recovery from surgery is required (Day 1 of Cycle 4 will be determined by the treating investigator once the subject is cleared to initiate systemic therapy). Nivolumab (480 mg IV infusion on Day 1 of each 4-week cycle) will be administered for up to 9 cycles during the Adjuvant phase.
  Interventions: Drug: Tavo; Drug: Nivolumab; Device: OncoSec Medical Electroporation Therapy System

INTERVENTIONS:
Drug: Tavo — Tavo will be injected on Days 1 and 8 every 4 weeks at a dose volume of ¼ of the calculated lesion volume with a minimum dose volume per lesion of 0.1 mL for lesions of volume <0.4 cm3
Drug: Nivolumab — Nivolumab will be administered 480 mg every 4 weeks over 30 minute infusions
Device: OncoSec Medical Electroporation Therapy System — The OMS (OncoSec Medical Electroporation Therapy System), a medical EP device system, consists of 3 components: 1. an Electroporation Generator that generates electric pulses, 2. a sterile Applicator Tip containing needle array, and 3. an Applicator Handle that connects to the Electroporation Generator at the proximal end and connects to the Applicator Tip at the distal end.
  Upon user activation of the attached Foot Switch, the OMS Electroporation Generator delivers controlled electrical pulses in a square wave pulse pattern yielding optimal transmembrane potential for electroporation to occur. EP pulses occur between 6 hexagonal opposing needle electrodes. After the first pulse, the polarity between the opposing needle electrode pairs is reversed and the needle pair is pulsed again. After the initial paired pulse, the pulse delivery is rotated clockwise to the next opposing needle pairs until a total of 6 pulses are delivered to complete the EP sequence.
  Other Names: Electroporation

SUMMARY:
This is a Phase 2 open-label, single-arm study of neoadjuvant treatment of intratumoral tavo-EP plus nivolumab IV infusion. Eligible participants will be those with pathological diagnosis of operable locally-regionally advanced melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥ 18 years of age inclusive, at the time of signing the informed consent
* Histologic diagnosis of melanoma
* Must be considered surgically operable and may present as any of the following groups:

  1. Primary melanoma with clinically apparent regional lymph node metastases, confirmed by pathological diagnosis.
  2. Clinically detected recurrence of melanoma at regional lymph node basin(s), confirmed by pathological diagnosis.
  3. Clinically or histologically detected primary melanoma involving multiple regional nodal groups, confirmed by pathological diagnosis.
  4. Clinically detected single site of nodal metastatic melanoma arising from an unknown primary, confirmed by pathological diagnosis.
  5. Participants with in transit or satellite metastases with or without lymph node involvement are allowed if they are considered surgically resectable at Screening by the treating surgical oncologist.
  6. Participants with distant cutaneous/subcutaneous, soft tissue or nodal metastases with or without regional lymph node involvement are allowed if they are considered potentially surgically resectable and can be biopsied at Screening by the treating surgical oncologist. Elevated LDH is not an exclusion.
* Participants are eligible for this study either at presentation for primary melanoma with concurrent regional nodal and/or in-transit or distant metastasis, or at the time of clinically detected nodal, in transit, or distant recurrence
* Participants must be evaluated by standard-of-care full body imaging studies including positron emission tomography - computed tomography (PET-CT ;preferred; including diagnostic CT component if possible) or CT (if PET-CT cannot be done) as well as magnetic resonance imaging (MRI) of the brain (or CT if MRI cannot be done) as part of the initial clinical work-up at Screening (no more than 4 weeks prior to Cycle 1, Day 1).
* Have measurable disease based on RECIST v1.1, with at least one anatomically distinct lesion. Lesion or lesions must meet all the following baseline criteria:

  1. Accessible for electroporation
  2. Must be measured in at least one dimension (longest diameter in the plane of measurement is to be recorded)
  3. Greater than 3 mm
* Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Male Participants: Male subjects of childbearing potential must be surgically sterile, or must agree to use adequate method of contraception during the study and at least 5 months following the last day of study drug administration. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject
* Female participants: Women of childbearing potential must have negative serum or urine pregnancy test within 72 hours prior to receiving the first study drug administration. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. For women of childbearing potential, must be willing to use an adequate method of contraception from 30 days prior to the first study drug administration and 5 months following last day study drug administration (either tavo or nivolumab); acceptable methods include hormonal contraception (oral contraceptives - as long as on stable dose, patch, implant, and injection), intrauterine devices, or double barrier methods (e.g. vaginal diaphragm/vaginal sponge plus condom, or condom plus spermicidal jelly), sexual abstinence or a vasectomized partner. Women may be surgically sterile or at least 1-year post-last menstrual period. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol

Exclusion Criteria:

* Participant has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer. Also, includes patients who are considered disease-free for at least 3 years from the last definitive treatment for a second malignancy.
* Participants who have Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies at Screening). HIV testing at screening is not required unless considered clinically indicated by the treating physician.
* Participants who have active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected at Screening); Note: Participants who have been vaccinated against Hepatitis B and who are positive only for the Hepatitis B surface antibody are permitted to participate in the study. Hepatitis B and C testing at screening is not required unless considered clinically indicated by the treating physician.
* Participant has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug. The use of physiologic doses of corticosteroids may be approved after consultation with the Principal Investigator.
* Participant has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Participant has a history of interstitial lung disease.
* Participant has an active infection requiring systemic therapy.
* Participant has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Participant has not recovered (i.e., > Grade 1 at Cycle 1, Day 1) from AEs due to a previously administered agent.
* Participant has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
* Participants who are pregnant or breast feeding or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 5 months after the last dose of trial treatment.
* Participants with electronic pacemakers or defibrillators
* Participants who have received a live-virus vaccination within 30 days of the first dose of treatment. Seasonal flu vaccines that do not contain live virus are permitted
* Participants who have received transfusion of blood products (including platelets or red blood cells) or administration of colony stimulating factors (including G-CSF, GM-CSF or recombinant erythropoietin) within 4 weeks prior to study Cycle 1, Day 1.
* Previous treatment with anti-PD1 or anti-PDL1 immunotherapy.
* Participation in another clinical study and systemic therapy within 30 days of Cycle 1, Day 1.
* ECOG Performance Status: >1
* Inadequate organ function as defined per protocol
* Participant has severe hypersensitivity (≥Grade 3) to nivolumab and/or any of its excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2024-03-26 (Actual); Study Completion 2028-06-15 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Tarhini, MD, PhD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Tarhini AA, Eroglu Z, Eljilany I, Zager JS, Gonzalez RJ, Sarnaik AA, Cruse CW, Khushalani NI, De Aquino DB, Abraham E, Acevedo DM, Richards A, Schell MJ, Kalos D, Chen PL, Messina JL, Canton DA, Sondak VK. Neoadjuvant Intratumoral Plasmid IL-12 Electro-Gene-Transfer and Nivolumab in Patients with Operable, Locoregionally Advanced Melanoma. Clin Cancer Res. 2024 Dec 2;30(23):5333-5341. doi: 10.1158/1078-0432.CCR-24-2768. PMID 39417680
- [Derived] Jacobs L, Yshii L, Junius S, Geukens N, Liston A, Hollevoet K, Declerck P. Intratumoral DNA-based delivery of checkpoint-inhibiting antibodies and interleukin 12 triggers T cell infiltration and anti-tumor response. Cancer Gene Ther. 2022 Jul;29(7):984-992. doi: 10.1038/s41417-021-00403-8. Epub 2021 Nov 9. PMID 34754076

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Neoadjuvant Treatment
Started | 17
Completed | 16
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Neoadjuvant Treatment
Number analyzed (Participants) | 16
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 69 [30 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response
Description: For each subject, the study intervention consists of 3 phases: (1) Neoadjuvant Phase; (2) Surgery Phase; (3) Adjuvant Phase. Completion of all 3 phases is required for primary completion of the study. The study protocol requires that all subjects will be followed for 4 weeks after last dose of nivolumab at End of Study (EOS) visit. That is 4 weeks after the conclusion of the adjuvant phase. For the purpose of reporting the primary outcome measure, Pathologic Complete Response will be estimated based on the proportion of participants who have completed the study phases and were found to have no viable tumor on histologic assessment at definitive surgery after the 12- week Neoadjuvant phase. Surgery will then be scheduled 2-4 weeks after neoadjuvant phase. This will be followed by the adjuvant phase. Therefore, the proportion of participants who continue in Pathologic Complete Response following completion of the 3 study phases would be reported.
Time Frame: At least four weeks after the last dose of nivolumab at End of Study (EOS) visit
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Treatment
Number analyzed (Participants) | 15
Participants | 9

2. Secondary Outcome: Objective Response Rate
Description: Preoperative ORR assessed by Investigator based on RECIST v1.1 at the conclusion of the Neoadjuvant phase.
Time Frame: Conclusion of the neoadjuvant phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Treatment
Number analyzed (Participants) | 16
Participants | 10

3. Secondary Outcome: Relapse Free Survival
Description: RFS assessed by Investigator based on RECIST v1.1 at least four weeks after the last dose of nivolumab at End of Study (EOS) visit.
Time Frame: At least four weeks after the last dose of nivolumab at End of Study (EOS) visit
Measure: Number (95% Confidence Interval); unit: 1-year RFS Probability
Arm/Group | Neoadjuvant Treatment
Number analyzed (Participants) | 16
1-year RFS Probability | 93 [80 to 100]

4. Secondary Outcome: Overall Survival
Description: Overall survival at 1 year after start of therapy.
Time Frame: At 1 year after start of therapy
Measure: Number (95% Confidence Interval); unit: 1 Year OS Percent Probability
Arm/Group | Neoadjuvant Treatment
Number analyzed (Participants) | 16
1 Year OS Percent Probability | 94 [83 to 100]

5. Secondary Outcome: Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]
Description: To determine the safety and tolerability of combined treatment as neoadjuvant therapy will be based on the frequency of AEs
Time Frame: Up to 5 years after start of therapy
Reporting Status: Not Posted

6. Secondary Outcome: Risk of Surgical Delay
Description: Definitive surgery will be planned at about 12 weeks. Participants will be monitored for surgical delay (either due to toxicity and/or tumor progression). Defined as the number of participants who had Surgery delayed due to progression.
Time Frame: Up to 16 weeks after start or therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Treatment
Number analyzed (Participants) | 16
Participants | 1

ADVERSE EVENTS:
Time Frame: 1 year
Description: Treatment Emergent: Related + Unrelated
Arm/Group | Neoadjuvant Treatment
All-Cause Mortality (participants affected / at risk) | 2/16
Serious Adverse Events (participants affected / at risk) | 8/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant Treatment (N=16)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Flu like symptoms (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant Treatment (N=16)
Hyperglycemia (Metabolism and nutrition disorders) | 9 (12)
Hyperkalemia (Metabolism and nutrition disorders) | 7 (13)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (5)
Hypoglycemia (Metabolism and nutrition disorders) | 4 (4)
Hyponatremia (Metabolism and nutrition disorders) | 4 (6)
Anorexia (Metabolism and nutrition disorders) | 3 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 (84)
Investigations - Other, specify (Investigations) | 5 (9)
Alkaline phosphatase increased (Investigations) | 4 (12)
Creatinine increased (Investigations) | 4 (5)
Aspartate aminotransferase increased (Investigations) | 3 (11)
INR increased (Investigations) | 3 (5)
Thyroid stimulating hormone increased (Investigations) | 3 (4)
Blood lactate dehydrogenase increased (Investigations) | 2 (2)
Lymphocyte count decreased (Investigations) | 2 (3)
Neutrophil count decreased (Investigations) | 2 (2)
Weight loss (Investigations) | 2 (3)
White blood cell decreased (Investigations) | 2 (3)
Alanine aminotransferase increased (Investigations) | 1 (3)
Platelet count decreased (Investigations) | 1 (2)
Fatigue (General disorders) | 9 (14)
Flu like symptoms (General disorders) | 3 (4)
Chills (General disorders) | 2 (2)
Edema limbs (General disorders) | 2 (2)
Pain (General disorders) | 2 (3)
Disease progression (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
Neck edema (General disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 7 (14)
Nausea (Gastrointestinal disorders) | 5 (8)
Constipation (Gastrointestinal disorders) | 4 (5)
Colitis (Gastrointestinal disorders) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 2 (3)
Bloating (Gastrointestinal disorders) | 1 (2)
Pancreatitis (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (3)
Dizziness (Nervous system disorders) | 5 (6)
Headache (Nervous system disorders) | 4 (7)
Ataxia (Nervous system disorders) | 1 (1)
Concentration impairment (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Vasovagal reaction (Nervous system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 8 (21)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 3 (3)
Upper respiratory infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Kidney infection (Infections and infestations) | 1 (1)
Pelvic infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Burn (Injury, poisoning and procedural complications) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (2)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (1)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1)
Agitation (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 1 (1)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 3 (4)
Myocardial infarction (Cardiac disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2 (2)
Renal calculi (Renal and urinary disorders) | 2 (2)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Hypertension (Vascular disorders) | 5 (10)
Hypotension (Vascular disorders) | 3 (4)
Lymphedema (Vascular disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (3)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Hypophysitis (Endocrine disorders) | 1 (1)
Hypopituitarism (Endocrine disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (2)
Eye disorders - Other, specify (Eye disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Immune system disorders - Other, specify (Immune system disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-26): https://cdn.clinicaltrials.gov/large-docs/30/NCT04526730/Prot_SAP_000.pdf